CLINICAL TRIAL: NCT02947009
Title: Exercise-induced Paradoxical Vocal Fold Motion Disorder: Clinical Feature Characteristics and Potential Mechanisms
Brief Title: Exercise-induced Paradoxical Vocal Fold Motion Disorder: Clinical Features and Potential Mechanisms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Adrianna Shembel, Principal Investigator, University of Pittsburgh
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1F31DC015752-01A1 (NIH)
Record Dates: First submitted 2016-10-19; First posted 2016-10-27 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2016-10

CONDITIONS: Disorder of Vocal Cord

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adolescent athletes with PVFMD (Experimental): participants must be adolescents (ages 12-18yo) who exercise regularly (at least 40 min 3x/week) and engage in athletic activities competitively by their report.
  Any participant who declares he or she is a competitive athlete and presents to the clinic reporting atypical dyspnea during exertion and associated decrements in athletic performance for more than 2 weeks prior to presentation will be considered for the study. Participants must score at least a 10 out of 40 on the Dyspnea Index
  Interventions: Behavioral: Diagnostic Study
- Adolescent athletes at-risk for PVFMD (Active Comparator): participants must be adolescents (ages 12-18yo) who exercise regularly (at least 40 min 3x/week) and engage in athletic activities competitively by their report.
  Participants in the at-risk group must report playing sports in a competitive environment, must report no symptoms of atypical dyspnea over the past 6 months, and must score less than 6 out of 40 on the Dyspnea Index.
  Interventions: Behavioral: Diagnostic Study

INTERVENTIONS:
Behavioral: Diagnostic Study — Participants will undergo laryngoscopy at baseline and with exercise challenge and will rate severity of various symptoms related to the larynx (ex. shortness of breath, voice changes, cough).

SUMMARY:
Exercise-induced paradoxical vocal fold motion disorder (E-PVFMD) - which severely impacts the lives of up to 1 million adolescents in the U.S. annually - is under- or mis-diagnosed in as many as 80% of cases, leading to ineffective, protracted periods of management. Additionally, what makes those with the condition different from those at risk for the condition (e.g., playing sports/engaging in athletic activity within a competitive athletic environment) is unclear. The goals of this proposed study are to address this diagnostic challenge by (1) pursuing a previously published preliminary taxonomic algorithm for the clinical identification and classification of EPVFMD, and by (2) elucidating potential underlying mechanisms driving this clinical presentation. Study outcomes will improve sensitivity and specificity of diagnosis protocols for PVFMD, thereby reducing prevalence of misdiagnosis and improving clinical management in individuals with this disorder in the future. Outcomes will also be used to create preventative care measures for adolescents at risk for the condition.

DETAILED DESCRIPTION:
The experimental protocol consists of five stages in total (Stages IV): (1) Screening, (2) Pre-Baseline, (3) Baseline Laryngoscopy Condition, (4) Exercise Laryngoscopy Condition, and (5) Recovery. The following sections describe procedures conducted within each of the five stages

Stage I: Screening

To determine eligibility, all consenting participants will (1) undergo spirometric screening to rule out any indication of pulmonary pathology, (2) report they partake in athletic activity within a competitive environment (self-perceived/reported), and (3) complete the Dyspnea Index (DI). Participants with less than 80% predicted FEV1 on spirometry will be excluded from the study and referred to the pediatric pulmonary clinic at Massachusetts General Hospital (MGH). Anyone who reports they feel their sports-related activities are not competitive will be excluded. Participants in the E-PVFMD group who score less than 10 out of 40 on the DI will be excluded from the study, whereas participants in the at-risk group who score more than 6 out of 40 on the DI will be excluded from the study.

Stage II: PreBaseline

All participants who have passed the screening will rate the worst severity of perceived shortness of breath experienced during the screening period, as well as other symptoms relating to PVFMD (i.e., cough, globus, dysphonia, laryngeal pain/tension), on a 0100mm visual analog scale (VAS). These values will later serve as anchors for subsequent symptom ratings. Rating severity of symptoms prior to laryngoscopy will also prime participants for symptom severity ratings in subsequent conditions, described shortly in detail. Next, blood pressure (SBP) and heart rate (HR) readings will be obtained three times (x3) at 30-second intervals or greater over a 5minute period, using a blood and heart rate monitor. The three readings will then be averaged and used as anchors for SBP and HR readings taken during subsequent study phases. Two self-reported questionnaires will then be administered to all enrolled participants: the Early Adolescent Temperament Questionnaire - Revised-short form (EATQ-R-SF) and the Paffenbarger Physical Activity Questionnaire (PPAQ). Participants will read and complete the two questionnaires on their own, although the PI or parent/guardian may clarify questions or help participants read instructions, especially with younger participants. Last, a respiratory transducer band will be placed on ribs 5-8 to measure respiratory rate (RR) and tidal volumes (TV). These parameters may be used to stratify/bin data, posthoc.

Stage III: Baseline Laryngoscopy Condition

Participants will be positioned upright in an examination chair and given a decongestant (e.g., Afrin®) in one nasal passage. The laryngeal vestibule will then be visualized with flexible nasoendoscopy (laryngoscopy) using halogen light. Subjects with structural or dynamic abnormalities occluding more than a third of the airway will be ruled out (and excluded, as needed) and normal laryngeal movement (i.e., abduction on inspiration and slight adduction on exhalation) will be confirmed at rest by both clinician and ENT physician. The laryngeal examination will then be recorded and glottic and supraglottic laryngeal configuration will be analyzed later offline. The PI will watch the participant's thoracic and abdominal cavity movement and will call the beginning of each inspiratory ("I") and expiratory ("E") phase as the participant breathes. The calls will be recorded on laryngeal examination videos and used to identify optimal periods within specific phases of the respiratory cycle from which to extract digital still images of the larynx. Participants will be asked to remain as relaxed as possible, but instructions will not relate to breathing so as not to bring attention to respiratory patterns. Three SBP and HR readings will be recorded for the second time with a blood pressure cuff every 30 seconds or more over a 5min period and averaged across the three trials. Once the endoscope has been removed, participants will be asked to rate perception of their worst severity of shortness of breath experienced during the baseline laryngoscopy condition on the 0-100mm VAS for the second time.

Stage IV: Exercise Laryngoscopy Condition

Participants will then undergo a graded exercise test (GXT) with cycle ergometer and simultaneous flexible laryngoscopy. The exercise challenge will parallel procedures in a previously described 1minute progressive incremental cycle ergometer protocol, starting at 50 watts (300 kgm/min), with increments of 50 watts every minute. Simultaneous laryngoscopic procedures, as well as SBP and HR recordings, will generally parallel those of the baseline laryngoscopic protocol in Stage III. To minimize risk of injury or overexertion, explicit instructions for the exercise protocol will be given to each participant prior to the start of the protocol. Once participants have communicated understanding, they will sit on the ergometer and the seat will be properly adjusted so there is a slight bend in the knee joint when the ball of the foot is on the pedal, with the pedal in its lowest position (~10-15° angle of knee flexion when the leg is extended). Once seated in position, participants will be instructed to relax the grip of the handlebar to prevent peripheral constriction, which could confound cardiovascular functions. The blood pressure cuff will be adjusted accordingly in the standard fashion and a pulse oximeter will be fitted on the participant's middle finger of the dominant hand to monitor oxyhemoglobin saturation during the exercise challenge. Participants will then be trained on rating perceived levels of exertion by pointing to the Borg Perceived Exertion Scale mounted on a board. The Borg scale goes from 6 to 20, where 6 represents no feelings of exertion and a score of 19 represents anaerobic activity that cannot be sustained for more than a minute. Borg severity ratings will be used to identify optimal level of exertion for measures extracted from video images during the exercise condition. During this task, participants will be encouraged not to vocalize and will be asked to rely solely on the board to communicate their perceived level of exertion for each incremental exercise load that will be imposed. The goal of this endeavor is to avoid movement of the vocal folds with vocalization, which may confound respiratory (non-phonatory) laryngeal configuration parameters. A head mount will then be placed on the participant's head and the head of the flexible endoscope will be inserted into the head mount, with the flexible camera dangling from the head mount below the head of the endoscope. Next, participants will be reminded of the Borg Scale ratings, and re-instructed as needed. For participants with potential E-PVFMD, instructions will also be provided to indicate induction of PVFMD attack with a "thumbs up" signal during the provocation challenge. All participants will be informed they will be encouraged to continue pedaling throughout the protocol until vigorous exercise levels are reached. Participants will also be reminded the protocol is voluntary and they can terminate the trial at any time. Once participants have communicated understanding and their willingness to continue, the flexible camera lens will once again be inserted into the same nostril, in the same manner as for the baseline laryngoscopy examination. Once the laryngeal vestibule has been identified with the laryngoscope, the flexible camera lens will then be secured to the ipsilateral nare with surgical tape to prevent movement of the scope in and out of the nose. The graded exercise test (GXT) will then begin at 50 watts (300 kgm/min) with target increases of 300 kgm/min every minute, per standard GXT protocol. Participants will be asked to maintain a 50-70 RPM pedal rate (displayed on the ergometer) with each incremental increase in load. For participants in the E-PVFMD group, incremental loads will continue until one of two events transpires: (1) E-PVFMD attack occurs (i.e., the participant experiences symptoms representative of previously experienced paroxysmal PVFMD episodes, and indicates induction of the episode with a "thumbs up" sign). Once the episode begins, videoendoscopy recordings will be obtained for an additional 30 seconds before the exercise laryngoscopy challenge is terminated, at which point the video recording will also be stopped. (2) No signs/symptoms of "attack" occur at the 3-minute mark with maximum exertion (19-20 Borg score), and the challenge is terminated. Results in these latter cases will be binned for future analysis beyond the scope of the proposed study. However, the sans-PVFMD-attack cohort in the PVFMD group will be excluded from analysis for the final n=25 in the present study and replaced until the targeted sample size (n = 25) has been reached. For the at-risk group, once a score of 19 on the Borg scale has been reported, 30 additional seconds of videoendoscopy will be recorded before the task is terminated. To terminate the protocol for both groups, the bike ergometer will first be reduced to 0 watts load and the laryngoscope will be removed from the nasopharynx. During the exertion task, SBP and HR will be recorded at the one minute mark, right before each additional incremental increase in load, and then again 1-2 times during maximum exertion (Borg scale 19-20) within the 30-second maximum exercise challenge (and subsequent videoendoscopic recording time frame). Participants will be on the bike a maximum of 10 minutes.

Stage V: Recovery

The cycle ergometer task will be stopped and SBP and HR will once again be recorded, this time at the 1-minute, 2-minute, and 3-minute post-max exertion time points, determined by a stopwatch. Participants will be asked to rate their worst perceived symptoms experienced during the exercise laryngoscopy task for the third (and final time) time using the 0-100 VAS. HR readings will then be used to calculate heart rate recovery (HRR) offline for further data analysis. Participants will then cycle for an additional 1-2 min for proper cool down to ensure cardiovascular parameters are back to baseline before they are helped off the bike.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents (ages 12-18yo)
* Exercise regularly (at least 40min 3x/week) in competitive athletic environment
* Inclusion criteria specific to E-PVFMD group: report of atypical dyspnea during exertion and associated decrements in athletic performance for more than 2 weeks prior to presentation; Score of > 10/40 on the Dyspnea Index

Exclusion Criteria:

* Developmental or cognitive disorder precluding ability to follow directions or read instructions
* Behavioral disorder that would disrupt study protocol or potentially affect outcome parameters (e.g., attention-deficit/hyperactivity disorder [ADHD], oppositional defiant disorder [ODD]).
* Neuromuscular disorders affecting the respiratory or phonatory system (e.g., ALS, Myasthenia Gravis)
* Supralaryngeal anatomical defects impeding airflow
* Cardiovascular conditions/disorders (e.g., hypertension)
* Poorly controlled obstructive pulmonary disorders (e.g., asthma)
* Use of the following medications: (a) antihypertensive, (b) cardiovascular, (c) psychotropic
* Identifiable (organic) vocal fold pathology occluding more than a 1/3 of the airway (e.g., lesions, nodules), found on laryngeal examination
* Intolerance to flexible nasoendoscopy
* E-PVFMD group only: absence of signs or symptoms of acute E-PVFMD attack with exercise provocation challenge at maximum exertion at or before the 3minute mark.
* At-Risk group only: Positive signs or symptoms of an acute E-PVFMD attack with exercise provocation challenge at maximum exertion.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2016-11; Primary Completion 2017-07-03 (Actual); Study Completion 2017-07-03 (Actual)

PRIMARY OUTCOMES:
Estimates of vocal fold angle at anterior commissure, determined on laryngoscopic digital images taken at height of inspiration prior to start of exhalation | 1 year
Self-report of dyspnea severity, determined on 100mm visual analog scale | 1 year

SECONDARY OUTCOMES:
Amount arytenoid prolapse, rated on a 0-3 scale based on videoendoscopic images | 1 year
Amount of epiglottic collapse, rated on a 0-3 scale based on videoendoscopic images | 1 year
Amount of ventricular compression, rated on a 0-3 scale based on videoendoscopic images | 1 year
Self-report of cough severity, determined based on 100mm visual analog scale | 1 year
Self-report of neck tightness severity, determined based on 100mm visual analog scale | 1 year
  self-reported ratings of symptoms of cough, globus sensation, neck tightness, dysphonia, and stridor
Self-report of stridor severity, determined based on 100mm visual analog scale | 1 year

OTHER OUTCOMES:
Estimates of autonomic balance, determined with systolic blood pressure at maximum exertion | 1 year
Estimates of autonomic balance, determined with heart rate recovery | 1 year
  Heart rate recovery determined by the difference between heart rate at maximum exertion and heart rate at the 2-minutes post-recovery time point.
Assessment of temperament, based on the Early-Adolescent Temperament Questionnaire - revised - short form (EATQ-R-SF) | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Mass Eye and Ear Infirmary, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abu-Hasan M, Tannous B, Weinberger M. Exercise-induced dyspnea in children and adolescents: if not asthma then what? Ann Allergy Asthma Immunol. 2005 Mar;94(3):366-71. doi: 10.1016/S1081-1206(10)60989-1. PMID 15801248
- [Background] Al-Alwan A, Kaminsky D. Vocal cord dysfunction in athletes: clinical presentation and review of the literature. Phys Sportsmed. 2012 May;40(2):22-7. doi: 10.3810/psm.2012.05.1961. PMID 22759602
- [Background] Altman KW, Mirza N, Ruiz C, Sataloff RT. Paradoxical vocal fold motion: presentation and treatment options. J Voice. 2000 Mar;14(1):99-103. doi: 10.1016/s0892-1997(00)80099-5. PMID 10764121
- [Background] Bittleman DB, Smith RJ, Weiler JM. Abnormal movement of the arytenoid region during exercise presenting as exercise-induced asthma in an adolescent athlete. Chest. 1994 Aug;106(2):615-6. doi: 10.1378/chest.106.2.615. PMID 7774352
- [Background] Carter JB, Banister EW, Blaber AP. Effect of endurance exercise on autonomic control of heart rate. Sports Med. 2003;33(1):33-46. doi: 10.2165/00007256-200333010-00003. PMID 12477376
- [Background] Christensen PM, Thomsen SF, Rasmussen N, Backer V. Exercise-induced laryngeal obstructions: prevalence and symptoms in the general public. Eur Arch Otorhinolaryngol. 2011 Sep;268(9):1313-9. doi: 10.1007/s00405-011-1612-0. Epub 2011 Apr 29. PMID 21528411
- [Background] Christopher KL, Morris MJ. Vocal cord dysfunction, paradoxic vocal fold motion, or laryngomalacia? Our understanding requires an interdisciplinary approach. Otolaryngol Clin North Am. 2010 Feb;43(1):43-66, viii. doi: 10.1016/j.otc.2009.12.002. PMID 20172256
- [Background] Coote JH. Recovery of heart rate following intense dynamic exercise. Exp Physiol. 2010 Mar;95(3):431-40. doi: 10.1113/expphysiol.2009.047548. Epub 2009 Oct 16. PMID 19837772
- [Background] Fahey JT, Bryant NJ, Karas D, Goldberg B, Destefano R, Gracco LC. Exercise-induced stridor due to abnormal movement of the arytenoid area: videoendoscopic diagnosis and characterization of the "at risk" group. Pediatr Pulmonol. 2005 Jan;39(1):51-5. doi: 10.1002/ppul.20076. PMID 15558600
- [Background] Gartner-Schmidt JL, Shembel AC, Zullo TG, Rosen CA. Development and validation of the Dyspnea Index (DI): a severity index for upper airway-related dyspnea. J Voice. 2014 Nov;28(6):775-82. doi: 10.1016/j.jvoice.2013.12.017. Epub 2014 Oct 12. PMID 25311596
- [Background] Johansson H, Norlander K, Berglund L, Janson C, Malinovschi A, Nordvall L, Nordang L, Emtner M. Prevalence of exercise-induced bronchoconstriction and exercise-induced laryngeal obstruction in a general adolescent population. Thorax. 2015 Jan;70(1):57-63. doi: 10.1136/thoraxjnl-2014-205738. Epub 2014 Nov 7. PMID 25380758
- [Background] Langdeau JB, Turcotte H, Desagne P, Jobin J, Boulet LP. Influence of sympatho-vagal balance on airway responsiveness in athletes. Eur J Appl Physiol. 2000 Nov;83(4 -5):370-5. doi: 10.1007/s004210000306. PMID 11138577
- [Background] Newman KB, Mason UG 3rd, Schmaling KB. Clinical features of vocal cord dysfunction. Am J Respir Crit Care Med. 1995 Oct;152(4 Pt 1):1382-6. doi: 10.1164/ajrccm.152.4.7551399.
- [Background] Noyes BE, Kemp JS. Vocal cord dysfunction in children. Paediatr Respir Rev. 2007 Jun;8(2):155-63. doi: 10.1016/j.prrv.2007.05.004. PMID 17574160
- [Background] Pierpont GL, Voth EJ. Assessing autonomic function by analysis of heart rate recovery from exercise in healthy subjects. Am J Cardiol. 2004 Jul 1;94(1):64-8. doi: 10.1016/j.amjcard.2004.03.032. PMID 15219511
- [Background] Roksund OD, Maat RC, Heimdal JH, Olofsson J, Skadberg BT, Halvorsen T. Exercise induced dyspnea in the young. Larynx as the bottleneck of the airways. Respir Med. 2009 Dec;103(12):1911-8. doi: 10.1016/j.rmed.2009.05.024. Epub 2009 Sep 26. PMID 19782550
- [Background] Shembel A, Kolouri S, Xu H, Verdolini Abbott K. Quantification of Respiratory Laryngeal Morphometry: Comparison of Laryngeal Lumen Angle Estimate Methods. J Voice. 2016 Nov;30(6):764.e23-764.e37. doi: 10.1016/j.jvoice.2015.10.011. Epub 2015 Dec 2. PMID 26652778
- [Background] Shembel AC, Sandage MJ, Verdolini Abbott K. Episodic Laryngeal Breathing Disorders: Literature Review and Proposal of Preliminary Theoretical Framework. J Voice. 2017 Jan;31(1):125.e7-125.e16. doi: 10.1016/j.jvoice.2015.11.027. Epub 2016 Feb 24. PMID 26922093
- [Background] Singh TP, Rhodes J, Gauvreau K. Determinants of heart rate recovery following exercise in children. Med Sci Sports Exerc. 2008 Apr;40(4):601-5. doi: 10.1249/MSS.0b013e3181621ec4. PMID 18317389
- [Background] Weinberger M, Abu-Hasan M. Perceptions and pathophysiology of dyspnea and exercise intolerance. Pediatr Clin North Am. 2009 Feb;56(1):33-48, ix. doi: 10.1016/j.pcl.2008.10.015. PMID 19135580
- [Background] Younes M, Burks J. Breathing pattern during and after exercise of different intensities. J Appl Physiol (1985). 1985 Sep;59(3):898-908. doi: 10.1152/jappl.1985.59.3.898. PMID 3932319